CLINICAL TRIAL: NCT05350774
Title: Immunotherapy for Neurological Post-Acute Sequelae of SARS-CoV-2 (IN-PASC)
Brief Title: Immunotherapy for Neurological Post-Acute Sequelae of SARS-CoV-2
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10000711; 000711-N
Record Dates: First submitted 2022-04-20; First posted 2022-04-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Systemic Inflammation; Neuroinflammation; Microvascular Thrombosis
Keywords: Long Haul Covid; COVID-19; Long Covid
MeSH Terms: conditions — Neuroinflammatory Diseases; Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Saline Solution; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVIg arm (Experimental): IVIg arm IV immunoglobulin 0.4g/kg/day for 5 days
  Interventions: Drug: IV immunoglobulin
- Placebo arm (Placebo Comparator): equivalent volume of Normal Saline for 5 days
  Interventions: Drug: IV normal saline

INTERVENTIONS:
Drug: IV normal saline — IV normal saline 250ml for 5 days
  Arms: Placebo arm
Drug: IV immunoglobulin — IVIg - IV immunoglobulin 0.4g/kg/day for 5 days
  Arms: IVIg arm

SUMMARY:
Background:

COVID-19 can cause problems in different parts of the body. For most people, it causes fevers or trouble breathing. Some people might not recover all the way. Researchers want to see if a treatment can help with people who have recovered from COVID-19 but still have symptoms ("Long COVID").

Objective:

To learn if human immunoglobulin (IVIG) will help with neurological symptoms of Long COVID.

Eligibility:

Adults ages 18 and older who had COVID-19 at least 12 weeks ago and have ongoing neurologic symptoms, such as dizziness, trouble walking, or problems with strength.

Design:

Participants will be screened with a medical record review.

Participants will have a medical history and a physical exam and complete questionnaires about their health and quality of life. They will have a spinal tap. They will give blood samples. They will discuss their symptoms with a neurologist and have a neurological exam.

Participants will take memory and thinking tests using a tablet. The tests will take 1 hour to complete. They will also take a smell and taste test. It will take approximately 30 minutes to complete.

Participants will lie on a table that tilts for up to 40 minutes. Their blood pressure and heart rate will be monitored. Blood will be taken through an intravenous (IV) catheter.

Participants will receive either IVIG, or saline by IV for 5 days. Then the participants will receive IVIG if they first received saline or saline if they first received IVIG by IV for another 5 days. They will not know what they receive.

Participants will have an MRI of the brain if they have not had one recently. They will receive a contrast agent by IV as part of the MRI scan.

Participants will be on the study for up to 4 months. They will have follow-up visits at the clinical center as well as fill out questionnaires at home. They may be asked to continue follow-up....

DETAILED DESCRIPTION:
Study Description:

This study will evaluate the clinical and laboratory effects of immunoglobulin therapy in patients who recovered from acute mild-moderate COVID-19 infection but still have persistent neurologic symptoms. Despite clinical recovery from the acute infection, some individuals continue to experience ongoing symptoms, at times several months after recovery, and many of these symptoms are neurologic. Some features suggest that this is a post-infectious immune-mediated process, and anecdotally patients have responded well to immunoglobulin therapy. This study will evaluate the clinical and laboratory effects of intravenous immunoglobulin therapy compared to placebo using a cross-over trial design. It is hypothesized that immunoglobulin therapy could have positive clinical and laboratory effects on patients with persistent neurological symptoms.

Objectives:

Primary Objective: To compare the clinical efficacy of intravenous immunoglobulin therapy to placebo in ameliorating the neurological post-acute sequalae of SARS-CoV-2 infection.

Secondary objective: To determine the clinical effects of intravenous immunoglobulin therapy in patients with neurological post-acute sequalae of SARS-CoV-2 infection.

Exploratory objective: To investigate the laboratory effects of intravenous immunoglobulin therapy in patients with neurological post-acute sequalae of SARS-CoV-2 infection.

Endpoints:

Primary endpoint:

Proportion of participants with a clinically meaningful change in Health Utilities Index Mark 3 (HUI3) 2 weeks after intravenous immunoglobulin therapy compared with 2 weeks after placebo.

Secondary endpoints:

* Change in functional / patient-reported scales:

  * WHO post COVID-19 functional scale
  * Post-COVID-19 Functional Status (PCFS) scale (0-4).
  * COVID-19 Yorkshire Rehabilitation Scale
  * PROMIS Global Health score
  * PROMIS Depression score
  * PROMIS anxiety score
* Change in clinical scales:

  * Montreal Cognitive Assessment (MoCA)
  * Brief tablet-based Neuropsychiatric evaluation
  * Karnofsky Performance Status (KPS)

Exploratory endpoints:

* Autonomic testing - Change in the number and character of test results indicating autonomic nervous system dysfunctions as evidenced by abnormal physiological responses to the Valsalva maneuver or head-up tilting.
* Change in immunological markers:

  * Cytokine levels
  * Cell markers per flow cytometry
  * SCENTinel, Olfactory testing, Monell

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged at least 18 and older.
* Meets the inclusion/exclusion criteria and is enrolled in Phase A of Protocol 000089 "Post-Coronavirus Disease 19 Convalescence at the National Institutes of Health."
* Previously diagnosed with mild-moderate COVID-19 (WHO Clinical Progression Scale between 2-5. Patients with severe acute COVID-19 requiring hospitalization or ICU care are excluded. Enrollment could take place 12 weeks after the diagnosis of acute COVID-19.
* Prior COVID-19 diagnosis confirmed by patient reported infection followed by confirmatory nucleocapsid antibody testing or a positive SARS-CoV-2 PCR test result from the time of infection.
* Exhibiting persistent neurologic symptoms evidenced by a self-reported illness narrative of the development of persistent PASC symptoms after recovering from a SARS-CoV-2 infection. These include symptoms such as fatigue, cognitive difficulties, orthostatic intolerance, and any ongoing issues with gait instability, vision, speech, swallowing, sensation or strength.
* Non-negligible PASC symptom severity, as determined using PCFS (minimal score of 2).
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Prior completion of a clinical brain MRI after the diagnosis of COVID-19, or willingness to complete a brain MRI.
* Meets current Clinical Center HES' policy for discontinuing isolation and quarantine for COVID-19.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

- For participants who have not completed a brain MRI since onset of symptoms: inability to complete brain MRI with gadolinium including contraindicated metal in the body, prior allergic reaction to gadolinium, eGFR <45 mmol/L, pregnancy or lactation, or claustrophobia that is unable to be adequately treated with a low dose oral

benzodiazepine.

* Contraindication to a research lumbar puncture, including use of anticoagulant medication, platelets < 50,000/uL, PT or PTT >1.5 x ULN for the NIH Clinical Center, or otherwise inability to complete the procedure.
* A condition that would significantly confound interpretation of the clinical and research tests as determined by the study investigators. This could include: traumatic brain injury, substance use disorder, active malignancy, systemic immunologic disorders, current or previous long-term immune suppressive therapy.
* Received a SARS-CoV-2 vaccine dose within less than 4 weeks of enrollment or is planning for any additional vaccines during the course of the study.
* Prior experimental treatment for PASC with immunoglobulins.
* Current medications include oral steroids or other immunosuppressive medications.
* Active participation in a clinical protocol which includes any intervention that may affect the results of the current study.
* Contraindication of intravenous immunoglobulins, including:

  * Renal insufficiency (eGFR<45mmol/L)
  * IgA deficiency
  * History of ischemic heart disease
  * Peripheral vascular disease
  * Cerebrovascular disease
  * Previously diagnosed hypercoagulability syndrome including antiphospholipid antibody syndrome, Protein C/S deficiency, Factor V Leiden, Antithrombin deficiency, MTHFR homozygosity
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 3.0 times the upper limit of normal.precluding the use of acetaminophen.
* Previously documented anaphylaxis or severe systemic reaction to immunoglobulins, acetaminophen, or diphenhydramine.
* A severe psychiatric condition, which based on the assessment of the study investigators, will impact the ability to complete the 12-week study course.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Effects of intravenous immunoglobulin therapy | 2 weeks
  Comparison of proportion of participants with a clinically meaningful change in Health Utilities Index Mark 3 (HUI3) after receiving either IVIg or placebo at Week 2.

SECONDARY OUTCOMES:
Investigate laboratory effects | 2 weeks
  Comparison of change in functional / patient-reported scales at 2 weeks after receiving each study intervention:a.<TAB>WHO post-COVID functional scale b.<TAB>PCFSc.<TAB>COVID-19 Yorkshire Rehabilitation Scaled.<TAB>PROMIS GHe.<TAB>PROMIS Depression f.<TAB>PROMIS Anxiety Comparison of change in clinical scales 2 weeks after receiving each study intervention:g.<TAB>Montreal Cognitive Assessment (MoCA)h.<TAB>Brief tablet-based Neuropsychiatric evaluation i.<TAB>Karnofsky Performance Status (KPS)

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000711-N.html